CLINICAL TRIAL: NCT03490357
Title: Quadratus Lumborum Versus Transversus Abdominis Plane Nerve Block: A Comparison in Regional Anesthesia Techniques With an Enhanced Recovery After Surgery Pathway
Brief Title: Quadratus Lumborum Versus Transversus Abdominis Plane Nerve Block: A Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00075597
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: The expected cephalad dermatomal distribution of the TAP block is T10. A positive outcome is a QL block with patient anesthesia at 2 or more dermatomes higher than the TAP block. The investigators will assume that there is a 30% difference between the two blocks, which leads to between 24 and 33 patients in each arm (ideally aiming for 30 patients in each group).
  The investigators have included other sample sizes should they find that there is a higher or lower percentage difference between the QL and TAP blocks.
  Outcome: A positive block is considered anesthesia at T8 or above and a negative block is considered analgesia below T8
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessor and patient blinded to type of block that the patient receives. Outcome assessor will check dermatomal levels after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Transversus Abdominus Plane Block (Active Comparator): Standardized ERAS regional nerve block
  Interventions: Procedure: Control - Transversus Abdominus Plane Block
- Quadratus Lumborum Block (Experimental): Quadratus lumborum nerve block
  Interventions: Procedure: Quadratus Lumborum Block

INTERVENTIONS:
Procedure: Control - Transversus Abdominus Plane Block — Abdominal fascial plane block - regional anesthesia
  Arms: Control - Transversus Abdominus Plane Block
Procedure: Quadratus Lumborum Block — Abdominal fascial plane block - regional anesthesia
  Arms: Quadratus Lumborum Block

SUMMARY:
The Transversus Abdominis Plane (TAP) block is the current standard of care for patients undergoing laparoscopic abdominal surgeries with the Enhanced Recovery After Surgery (ERAS) Protocol. The Quadratus Lumborum (QL) is another established abdominal fascial plane block that is comparable in procedure and risks and may potentially be more beneficial. The study compares the two blocks in hopes of establishing a new standard of care for patients undergoing laparoscopic abdominal surgeries with the ERAS protocol.

DETAILED DESCRIPTION:
The Transversus Abdominis Plane (TAP) block is the current standard of care for patients undergoing laparoscopic abdominal surgeries with the Enhanced Recovery After Surgery (ERAS) Protocol. The Quadratus Lumborum (QL) is another established abdominal fascial plane block that is comparable in procedure and risks and may potentially be more beneficial. The study compares the two blocks in hopes of establishing a new standard of care for patients undergoing laparoscopic abdominal surgeries with the ERAS protocol.

* Compare QL and TAP blocks cephalad spread via mapping in the Postoperative Acute Care Unit (PACU) within 6 hours after block placement.
* Compare efficacy of blocks via Visual Analogue Scale (VAS) pain scores in PACU and postoperative day (POD) 1.
* Compare amount of opioid pain medications consumed within 24 hours after block. Hypothesis
* The QL block will prove superior to the TAP block in both cephalad spread and pain control for abdominal surgery patients and decrease the amount of opioid pain medications required while in effect up to 24 hours after surgery.
* The quadratus lumborum will have increased cephalad spread. We predict mapping will show greater (2 or more dermatomal levels) or equal analgesic coverage by the QL block when compared to the TAP block.

ELIGIBILITY:
Inclusion Criteria:

* • Patients scheduled for laparoscopic abdominal surgery as posted by the surgeon

  * Part of the ERAS protocol as listed by the surgeon
  * Age 18 years and older
  * Elective procedure

Exclusion Criteria:

* • Patient inability to consent

  * Patient inability to communicate for data collection
  * Conversion from laparoscopic to open case
  * Local anesthetic allergy
  * Weight less than 50 kg
  * Anatomical variation making block visualization unlikely
  * Inability to cooperate with block
  * Surgery posted longer than 6 hours
  * Known preoperative substance abuse
  * Chronic opioid use > 3 months
  * Patient exhibits dependence on opioids Daily opioid use for pain control

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Dermatomal Mapping | 6 hours
  The primary outcome of interest is the proportion of subjects reporting a positive block. This is determined by dermatomal mapping in cephalad direction in PACU within 6 hours of TAP or QL placement. A positive outcome is one where the QL block measures 2 or more dermatomal levels higher than the TAP block

CONTACTS AND LOCATIONS:
Overall Officials: Renuka M George, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- The Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] George RM, McSwain JR, Gukasov M, Wilson DA, Nitchie H, Wilson SH. Dermatomal spread in lateral quadratus lumborum blocks versus transversus abdominus plane blocks after laparoscopic colorectal surgery: a randomized clinical trial. Reg Anesth Pain Med. 2024 Nov 7:rapm-2024-105488. doi: 10.1136/rapm-2024-105488. Online ahead of print. PMID 39510803